CLINICAL TRIAL: NCT06004141
Title: Pilot Randomized Controlled Trial of an Artificial Intelligence (AI)-Powered Behavioral Coaching Intervention (Laguna Health) to Promote Post-Hospital Discharge Recovery for Patients With Cancer
Brief Title: Behavioral Coaching Intervention (Laguna Health) for Patients With Cancer
Acronym: LAGUNA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to withdrawal of funding from Sponsor (Laguna Health)
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Laguna Health, Inc (Industry)
Responsible Party: Principal Investigator, Tejaswini M. Dhawale, MD, Instructor in Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-358
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Cancer
Keywords: Transitions of care; Hospitalization; Quality of Life; Behavioral Coaching; Home care; Neoplasm; Supportive Care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laguna Health Group (Experimental): * Patient and caregiver participants will have access to Laguna Health coaching and the Laguna Health mobile platform for 12 weeks after discharge from the hospital to a home environment.
  * Patient participants will receive usual post-discharge care as arranged by their inpatient and outpatient oncology teams.
  * Patient participants will complete study questionnaires to assess their quality of life, symptoms, and psychological outcomes.
  * Caregiver participants will complete study questionnaires to assess their quality of life and caregiving burden.
  * 10-20 participants will complete exit interviews to ascertain more feedback on the Laguna Health intervention.
  Interventions: Behavioral: Laguna Health
- Usual Care (No Intervention): * Participants will receive usual post-hospital discharge care as arranged by their inpatient and outpatient oncology care teams.
  * Patient participants will complete study questionnaires to assess their quality of life, symptoms, and psychological outcomes.
  * Caregiver participants will complete study questionnaires to assess their quality of life and caregiving burden.

INTERVENTIONS:
Behavioral: Laguna Health — Laguna Health is a novel behavioral coaching intervention (Laguna Health) that provides supportive care to patients with cancer who are discharged from the hospital and their caregivers. The intervention includes four components: 1) behavioral coaching with a Laguna Health recovery coach; 2) digital psycho-educational content tailored to the needs of patients with cancer; 3) summary of post-discharge care tasks; and 4) behavioral strategies to promote self-efficacy.
  Arms: Laguna Health Group

SUMMARY:
The overall goal of this study is to examine the feasibility, acceptability, and preliminary efficacy of using a behavioral coaching intervention (Laguna Health) for optimizing post-hospital discharge care in patients with cancer. Patients will be randomly assigned into one of the study groups: the behavioral coaching intervention (Laguna Health) + usual care versus usual care alone.

The Laguna Health intervention has several components:

1. Post-Discharge Recovery Coaching with a Laguna Health recovery coach to help patients identify barriers to post-discharge recovery
2. Digital psycho-educational content tailored to the needs of patients with cancer
3. Personal healthcare summaries
4. Digital content and coaching on behavioral strategies to promote self-efficacy

DETAILED DESCRIPTION:
This is a single-center, randomized, controlled research study to test the feasibility, acceptability and preliminary efficacy of Laguna Health for improving post-hospital discharge care in patients with cancer.

Laguna Health is behavioral coaching intervention wherein patients and their caregivers are paired with a Laguna Health recovery coach to promote post-discharge recovery. Additionally, Laguna Health offers patients and their caregivers access to a mobile platform containing psycho-educational content, healthcare summaries, and interactive features such as journaling and task lists.

Participants will be randomized in 1:1 fashion to one of the two study groups: Laguna Health + usual care versus usual care alone, stratified by cancer type and therapy intent (curable solid tumor vs. incurable GI cancer vs. incurable other solid tumor vs hematologic malignancy).

Participants randomly assigned to the Laguna Health group will receive access to the Laguna Health recovery coach and mobile platform for 12 weeks after they are discharged from the hospital.

Participants randomly assigned to the usual care group will receive usual post-hospital discharge care as arranged by their inpatient oncology team. They will not be given access to the Laguna Health intervention.

In both groups, participants are asked to complete questionnaires at baseline, weeks 6, weeks 12 and weeks 24 after enrolling in the study.

It is expected that 80 patients and at most 80 caregivers will take part in this study.

Laguna Health, Inc. is supporting this research study by providing funding.

ELIGIBILITY:
Inclusion Criteria (Patients):

* Adult patients (age > 18 years)
* Patients with cancer being treated with curative intent per chemotherapy order entry, treatment intent designation and or trial consent forms OR based on documentation in the oncology clinic notes.
* Patients with cancer being treated with palliative intent (per chemotherapy order entry, treatment intent designation and or trial consent forms OR based on documentation in the oncology clinic notes for those not receiving chemotherapy) who are experiencing their first or second hospitalization for cancer related care or complications.
* Unplanned or non-elective hospitalization at Massachusetts General Hospital (MGH)
* Planned discharge to a home environment.
* Receiving outpatient care at the MGH Cancer Center
* Access to a smartphone capable of accessing Laguna Health's app on Android or iOS
* Ability to comprehend, read, and respond to questions in English.

Exclusion Criteria (Patients):

* Patients with metastatic or advanced cancer experiencing their third or later hospitalization for cancer related care or complications as these patients likely have advanced disease and require more end-of-life care interventions.
* Patients with planned discharge to hospice or care facility other than home.
* Patients with acute or unstable psychiatric or cognitive conditions which the treating clinicians believes prohibits informed consent or compliance with study procedures

Caregiver Eligibility

* Adult (> 18 years) relative or friend of a patient who agrees to participate in the study whom the patient identified as living with them or having in-person contact with them at least twice per week.
* Ability to comprehend, read, and respond to questions in English as Laguna Health is only available in English in this proof-of-concept study.
* Access to a smartphone capable of accessing Laguna Health's app on Android or iOS

Note that patients can enroll without an eligible caregiver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Feasibility of Laguna Health based on enrollment and intervention use rates | Baseline to week-2
  Laguna Health will be deemed feasible if at least 60% of eligible patients are enrolled in the study, and of those patients enrolled and randomized to the intervention arm, 60% engage with the Laguna Health platform during at least 7 weeks of the 12-week post discharge intervention period.

SECONDARY OUTCOMES:
Acceptability of Laguna Health for patients with cancer who are discharged from the hospital | Week-12
  Laguna health will be acceptable to patients, defined by at least 80% of patients reporting satisfaction (score > 20, corresponding to scale midpoint) on the 8-item Client Satisfaction Questionnaire (CSQ-8). Total scores on the CSQ-8 range from 8 to 32 with the higher number indicating greater satisfaction.
Acceptability of Laguna Health for caregivers of patients patients with cancer who are discharged from the hospital | Week-12
  Laguna health will be acceptable to caregivers, defined by at least 80% of caregivers receiving Laguna reporting satisfaction (score > 20, corresponding to scale midpoint) on the 8-item Client Satisfaction Questionnaire (CSQ-8). Total scores on the CSQ-8 range from 8 to 32 with the higher number indicating greater satisfaction.
Patient Quality of Life (QOL) (FACT-G) | Baseline to week-24
  Compare patient QOL as assessed by the Functional Assessment of Cancer Therapy -General (FACT-G) between the two study groups longitudinally. The FACT-G is a 27-item QOL measure that assesses physical, social, emotional, and functional wellbeing during the prior seven days. Scores range from 0-108, with higher scores indicating better QOL.
Patient symptom burden (ESAS-R) | Baseline to week-24
  Compare patient symptom burden, as assessed by the Edmonton Symptom Assessment Scale (ESAS-R) between the two study groups. The ESAS-R is a 10-item measure that assesses various symptoms relevant to patients with cancer. The ESAS-R score range 0-100 with higher scores indicating worse symptom burden.
Patient anxiety symptoms (HADS-Anxiety subscale) | Baseline to week-24
  Compare anxiety symptoms, as assessed by the self-reported Hospital Anxiety and Depression Scale (HADS), between the study groups. The HADS is a 14-item measure with subscales to evaluate symptoms of anxiety and depression. The HADS consists of two subscales assessing depression and anxiety symptoms, with scores ranging from 0 (no distress) to 21 (maximum distress) with higher scores indicating worse anxiety symptoms.
Patient depression symptoms (HADS-Depression subscale) | Baseline to week-24
  Compare depression symptoms, as assessed by the self-reported Hospital Anxiety and Depression Scale (HADS) between the study groups. The HADS is a 14-item measure with subscales to evaluate symptoms of anxiety and depression. The HADS consists of two subscales assessing depression and anxiety symptoms, with scores ranging from 0 (no distress) to 21 (maximum distress) with high scores indicating worse depression symptoms.
Patient Post-Traumatic Stress Disorder (PTSD) (PCL) | Baseline to week-24
  Compare post-traumatic stress symptoms as assessed through the Post-traumatic Stress Disorder Checklist-Civilian Version between the study groups. The PCL is a 17-item PTSD Checklist that evaluates severity of PTSD symptoms. Scores range from 17-85 with higher scores indicating worse PTSD symptoms

OTHER OUTCOMES:
Patient self-efficacy (CASE) | Baseline to week-24
  Compare patient self-efficacy, as assessed through the Cancer Self-Efficacy Scale (CASE) between the study groups. The CASE is a commonly utilized measure to assess patients' confidence in managing the impact of their illness. This is a 17-item questionnaire with higher scores (range = 0-170) indicating higher levels of self-efficacy.
Caregiver Quality of Life (CarGOQOL) | Baseline to week-24
  Compare caregiver QOL as assessed through the Caregiver Oncology Quality of Life Questionnaire (CarGOQoL) between the study groups. The CARGOQOL is a validated measure of caregiver QOL. The CARGOQOL ranges from 0-100 with higher scores indicating better QOL.
Caregiving burden (CRA) | Baseline to week-24
  Compare caregiving burden as assessed through the Caregiver Reaction Assessment (CRA) between the two study groups. The CRA ranges from 24-120 with higher scores indicating greater caregiving burden.
Health Care Utilization | up to week 24
  Electronic Health Records (EHR) will be used to assess patient health care utilization including days alive and out of hospital, unplanned readmissions, post-discharge appointment attendance, and emergency department visits during the first 12 and 24 weeks after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Tejaswini Dhawale, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Tejaswini Dhawale, MD. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation
URL: http://www.partners.org/innovation